CLINICAL TRIAL: NCT04369391
Title: A Randomized, Single-dose, Crossover Study of the Effects of SEP-363856 on Electrocardiogram (ECG) Intervals in Subjects With Schizophrenia
Brief Title: A Clinical Study to Investigate the Effect of an Investigational Drug on Electrocardiogram Intervals in Adults With Schizophrenia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SEP361-114
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized using a double Williams design in equal ratio to six possible sequences of receiving the three treatments being studied:
  SEP-363856 150mg, Matched Placebo, moxifloxacin 400mg.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEP363856 150 mg (Experimental): SEP363856 tablet 150 mg
  Interventions: Drug: SEP363856 150 mg
- Placebo (Placebo Comparator): matched placebo
  Interventions: Drug: Placebo
- moxifloxacin 400 mg (Active Comparator): moxifloxacin tablet 400 mg
  Interventions: Drug: moxifloxacin 400 mg

INTERVENTIONS:
Drug: SEP363856 150 mg — SEP363856 tablet 150 mg
  Arms: SEP363856 150 mg
Drug: Placebo — Placebo tablet
  Arms: Placebo
Drug: moxifloxacin 400 mg — moxifloxacin tablet 400 mg
  Arms: moxifloxacin 400 mg

SUMMARY:
A clinical study to investigate the effect of an investigational drug in adults with schizophrenia by using Electrocardiogram (Picture of the electrical action of the heart). This study is accepting male and female participants between 18 years old -65 years old who have been diagnosed with schizophrenia. This study will be conducted in approximately 7 locations in the US. The study will last approximately 7 weeks.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, single-dose, active and placebo controlled, 3-period crossover study of the effect of SEP-363856 150 mg on electrocardiogram (ECG) intervals in subjects with schizophrenia. SEP-363856 and matching placebo will be utilized in a double-blind fashion. Moxifloxacin will be utilized as an active control in an open-label fashion.

The primary analysis will be based on concentration-QTc modeling of the relationship between plasma concentrations of SEP-363856 or its metabolite SEP-363854 and change-from baseline QTc.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 65 years of age, inclusive, at the time of informed consent
* Subject must give written informed consent and privacy authorization prior to participation in the study
* Subject meets DSM-5 criteria for a primary diagnosis of schizophrenia as established by clinical interview
* Subject must have a CGI S score ≤ 4 at Screening
* Subject must have a PANSS total score ≤ 80 at Screening
* Subject must have a score of ≤ 4 on the following PANSS items at Screening:

  * P7 (hostility)
  * G8 (uncooperativeness)
* Subject must have normal to mild symptoms on all individual items of the SAS (< 2), AIMS (< 3) and BARS (< 3) at Screening
* Subject must be clinically stable for the past three months in the opinion of the Investigator
* Subject has been taking an antipsychotic for at least six weeks prior to Screening and has had no change in antipsychotic medication(s) for at least six weeks prior to Screening
* Subject is, in the opinion of the Investigator, generally healthy based on Screening medical history, physical examination, neurological examination, vital sign measurement, electrocardiogram and clinical laboratory values

Exclusion Criteria:

* Subject has a DSM 5 diagnosis or presence of symptoms consistent with a DSM 5 diagnosis other than schizophrenia. Exclusionary disorders include but are not limited to alcohol use disorder (within past 12 months), substance (other than nicotine or caffeine) use disorder within past 12 months, major depressive disorder, bipolar I or II disorder, schizoaffective disorder, obsessive compulsive disorder and posttraumatic stress disorder. Symptoms of mild to moderate mood dysphoria or anxiety are allowed so long as these symptoms are not the primary focus of treatment
* Subject tests positive for drugs of abuse or alcohol at Screening
* Subject is at significant risk of harming him/herself or others (passive or active) according to the Investigator's judgment.
* Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study
* Female subject who is pregnant or lactating
* Subject has any clinically significant abnormal laboratory value(s) at Screening as judged by the Investigator
* Subject has an abnormal, clinically significant 12-lead ECG at screening
* Subject has experienced significant blood loss (≥ 473 mL) or donated blood within 60 days prior to first dose of study drug; has donated plasma within 72 hours prior to the first dose of study drug or intends to donate plasma or blood or undergo elective surgery during study participation or within 60 days after the last study visit.
* Subject has an abnormal, clinically significant 12-lead ECG at screening
* Subject has a history of sick sinus syndrome, first, second, or third-degree AV block,myocardial infarction, NYHA Class II-IV heart failure, cardiomyopathy, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, congenital long QT syndrome, family history of long QT, or moderate to severe hypokalemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Placebo-adjusted change-from-baseline QTc interval (ΔΔQTc) | 24 Hours

SECONDARY OUTCOMES:
Change from baseline in heart rate, QTcF, pulse rate, and QRS intervals (∆HR, ΔQTcF, ΔPR, and ∆QRS) | 24 Hours
If a substantial heart rate (HR) effect is observed: Change from baseline in QTcS, QTcI, and QTcP (ΔQTcS, ΔQTcI, and ΔQTcP) | 24 Hours
Placebo-adjusted change from baseline in heart rate, pulse rate, and QRS intervals (ΔΔHR, ΔΔPR, and ΔΔQRS) | 24 Hours
If a substantial heart rate (HR) effect is observed: Placebo-adjusted ΔQTcS, and/or ΔQTcI, and/or ΔQTcP, and/or ΔQTcF (ΔΔQTcS, ΔΔQTcI, ΔΔQTcP, ΔΔQTcF) if not selected as the primary endpoint | 24 Hours
Categorical summary for QTcF, heart rate, pulse rate, and QRS intervals | 24 Hours
If a substantial heart rate (HR) effect is observed: Categorical summary for QTcS, QTcI, and QTcP | 24 Hours
Frequency of treatment-emergent changes of T-wave morphology and U-waves presence. | 24 Hours

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Woodland International Research Group, Little Rock, Arkansas
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - California Neuropsychopharmacology Clinical Research Institute-LA, LLC (CNRI-LA, LLC), Pico Rivera, California
  - California Neuropsychopharmacology Clinical Research Institute-San Diego, LLC (CNRI-SD, LLC), San Diego, California
  - Research Centers of America, LLC, Hollywood, Florida
  - Hassman Research Institute, Marlton, New Jersey
  - Community Clinical Research Inc. Austin, TX 78754, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com